CLINICAL TRIAL: NCT01770704
Title: Chinese Observation Study of the Clinical Management of Bipolar Disorder
Brief Title: Observation Study of the Clinical Management of Bipolar Disorder
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: NIS-NCN-XXX-2012/1
Record Dates: First submitted 2013-01-16; First posted 2013-01-18 (Estimated); Last update posted 2016-04-07 (Estimated); Status verified 2016-04

CONDITIONS: Bipolar Disorder
Keywords: Bipolar disorder; Clinical management; Clinical outcomes
MeSH Terms: conditions — Bipolar Disorder

STUDY DESIGN:
Observational Model: Cohort
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients diagnosed with bipolar disorder I or II

SUMMARY:
The objective of the ambispective cohort study is to describe clinical management and clinical outcomes related to bipolar disorder in China, and establish the factors associated with different management patterns and clinical outcomes, provide psychiatrists with reliable and up-to-date information on the disease.

ELIGIBILITY:
Inclusion Criteria:

* Provision of subject informed consent.
* Diagnosis of Bipolar Disorder I or II (DSM-IV TR) in any phase of the disorder.
* Patients who had at least one mood event( depression, mania, hypomania or mixed) according to DSM-IV TR definition during the 3 and 12 months prior to the beginning of the study.

Exclusion Criteria:

* Inability to complete Patient Reported Outcomes (PROs) questionnaires.
* Participation in an interventional clinical study in last 12 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with bipolar disorder I or II with at least one mood event during the 3 and 12 months prior to the beginning of the study.
Sampling Method: Probability Sample
Enrollment: 520 (Actual)
Dates: Start 2013-02; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Number of episodes (depression, mania, hypomania or mixed). | Up to 21 months

SECONDARY OUTCOMES:
Treatments received for Bipolar Disorder: medication time. | Up to 21 months
Treatments received for Bipolar Disorder: medication classes. | Up to 21 months

CONTACTS AND LOCATIONS:
Overall Officials: Yu Xin, Principal Investigator — Beijing No.6 Hospital; Wang Gang, Principal Investigator — Capital Medical University
Locations (6):
- China (6):
  - Research Site, Beijing, Beijing Municipality
  - Research Site, Shenzhen, Guangdong
  - Reserach Site, Shanghai, Shanghai Municipality
  - Research Site, Xi’an, Shanxi
  - Research SIte, Kunming, Yunnan
  - Research Site, Hangzhou, Zhejiang

REFERENCES:
- [Derived] Xu JJ, Zhu XQ, Liu S, Ding LY, Fu BB, Sun CC, Pan YL, Wang W, Zhang L. Sociodemographic, clinical and treatment characteristics of current rapid-cycling bipolar disorder: a multicenter Chinese study. Int J Bipolar Disord. 2024 Apr 9;12(1):11. doi: 10.1186/s40345-024-00332-z. PMID 38592605
- [Derived] Shi X, Zhao Y, Yang H, Xu X, Fang Y, Yu X, Tan Q, Li H, Sun G, Wu H, Wang P, Yang J, Zhu X, Wang G, Zhang L. Factors associated with hospitalization times and length of stay in patients with bipolar disorder. Front Psychiatry. 2023 May 19;14:1140908. doi: 10.3389/fpsyt.2023.1140908. eCollection 2023. PMID 37275983
- [Derived] Zhang ZF, Huang J, Zhu XQ, Yu X, Yang HC, Xu XF, Fang YR, Tan QR, Li HC, Wang G, Zhang L. Clinicodemographic correlates of psychotic features in bipolar disorder - a multicenter study in China. BMC Psychiatry. 2023 May 24;23(1):365. doi: 10.1186/s12888-023-04761-5. PMID 37226150
- [Derived] Zhang L, Yang HC, Xu XF, Fang YR, Yu X, Tan QR, Li HC, Ungvari GS, Ng CH, Wang G, Xiang YT. Demographic and clinical differences between early- and late-onset bipolar disorders in a multicenter study in China. Psychiatry Res. 2016 Dec 30;246:688-691. doi: 10.1016/j.psychres.2016.10.063. Epub 2016 Oct 30. PMID 27825780
- See also: NIS-NCN-XXX-2012_1-Bipolar Disorder in China_NISR_20151126 CSR Synopsis — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=907&filename=NIS-NCN-XXX-2012_1-Bipolar%20Disorder%20in%20China_NISR_20151126-CSR%20SYNOPSIS.pdf